CLINICAL TRIAL: NCT05582681
Title: HCV Test and Treat Utilizing Simplified HCV Patient Education
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The funding was halted.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-06023705
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Hepatitis C
Keywords: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Intervention Model Description: This is an open label, phase 4 randomized trial to assess test and treat strategy with simplified video-based patient education versus standard of care referral with health care provider delivered patient education.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HCV Education (Active Comparator): The intervention of HCV education will be performed at the addiction care setting for video- based patient education. Health care provide delivered patient education is the standard of care referral approach. HCV Education will include HCV disease overview, HCV screening, taking Glecaprevir/Pibrentasivir (G/P), and post study drug assessment and management. Participants may be randomized to either the video-based patient education or the HCV delivered patient education.
  Interventions: Other: HCV education from a health care provider; Drug: Glecaprevir and Pibrentasvir
- Point of Care (POC) HCV Viremia (RNA) testing (Experimental): All participants will have standardized laboratory assessments for HCV Viremia (RNA testing) as well as Cepheid POC HCV Viremia (RNA) test. The Cepheid Xpert HCV Viral Load (VL) Fingerstick assay is a test designed for the quantitation (amount) of Hepatitis C Virus (HCV) DNA in human whole blood. The HCV RNA result will be compared to standardized laboratory assessment for HCV Viremia. The Cepheid test is being conducted for research use only and will not be used for HCV diagnosis or treatment decisions.
  Interventions: Diagnostic Test: Cepheid POC HCV Viremia (RNA) test; Other: HCV education from a health care provider; Drug: Glecaprevir and Pibrentasvir

INTERVENTIONS:
Diagnostic Test: Cepheid POC HCV Viremia (RNA) test — The Cepheid Xpert HCV Viral Load (VL) Fingerstick assay is a test designed for the quantitation (amount) of Hepatitis C Virus (HCV) DNA in human whole blood. The HCV RNA result will be compared to standardized laboratory assessment for HCV Viremia. The Cepheid test is for being conducted for research use only and will not be used for HCV diagnosis or treatment decisions.
  Arms: Point of Care (POC) HCV Viremia (RNA) testing
Other: HCV education from a health care provider — HCV education provided by health care provider. HCV Education will include HCV disease overview, HCV screening, treatment with G/P, and post treatment assessment and management
Drug: Glecaprevir and Pibrentasvir — G/P will be provided for 8 weeks.
  Other Names: G/P

SUMMARY:
The study hypothesis is that the test and treat model utilizing video-based patient education will have higher rates of hepatitis C virus (HCV) treatment initiation and treatment completion.

DETAILED DESCRIPTION:
Viral hepatitis C (HCV) represents a major public health concern and is associated with significant morbidity and mortality. HCV screening and treatment among people who use drugs is challenging due to barriers leading to loss within HCV care cascades at most centers providing addiction care.

One critical element that would improve access to HCV therapy would be a test, educate and treat system, where people obtain drug on the same day as they are confirmed as Hepatitis C viremic.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age greater or equal to18 at study entry or emancipated minors over greater or equal to 16 to less or equal 70 years at study entry
* HCV antibody positive
* HCV treatment naïve (no prior treatment with an approved or investigational anti HCV medication)

Exclusion Criteria:

* Current or history of decompensated liver disease (including but not limited to encephalopathy, variceal bleeding, or ascites) prior to study entry
* History of hepatocellular carcinoma (HCC)
* Any history of active Hepatitis B or positive HBsAg positive test
* HCV RNA undetectable

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Number of subjects who initiated treatment within 8-week window from enrollment. | Up to 8 weeks

SECONDARY OUTCOMES:
Number of subjects who complete treatment in 8 weeks | Up to 8 weeks
Sustained Viral Response 12 weeks post dosing (SVR12) (<lower limit of quantification (LLOQ) of HCV RNA in at 12 weeks post treatment with window up to 24 weeks after end of treatment) | Up to 24 weeks
SVR12 (<LLOQ of HCV RNA in at 12 weeks post treatment with window up to 24 weeks after end of treatment) from real world evidence post-marketing observational study (RWE PMOS) efficacy G/P9 (compare test and treat arm with PMOS SVR12 result) | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Brown, MD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Phoenix House, Long Island City, New York
  - ColumbiaDoctors Midtown, New York, New York
  - Weill Cornell Medicine Midtown Center for Treatment and Research, New York, New York

IPD SHARING:
Plan to Share IPD: No